## INFORMED CONSENT "LET'S TALK ABOUT COLLEGE STUDENT SLEEP: AN INNOVATIVE NON-INVASIVE NEUROMODULATION TREATMENT TO IMPROVE SLEEP QUALITY AND ACADEMIC PERFORMANCE: RANDOMIZED CLINICAL TRIAL" (USLEEP)

**ID: USLEEP** 

[NCT ID not yet assigned] 15/11/2021



"Let's Talk About College Student Sleep: An Innovative Non-invasive Neuromodulation Treatment to Improve Sleep Quality and Academic Performance: Randomized Clinical Trial" (USLEEP)

## Informed consent

This consent form is aimed at FIRST-YEAR PHYSIOTHERAPY STUDENTS who are going to participate in the study "Let's talk about sleep in university students: an innovative non-invasive neuromodulation treatment to improve sleep quality and academic performance: Clinical trial randomized ".

This research is conducted by Dr. Pablo Aparicio Montero from the Alfonso X el Sabio University of Madrid, Dr. Raquel Medina from the University of Las Palmas de Gran Canaria, Dr. Alberto Meilán, from the Pontifical University of Salamanca and Dr. Daniel Pecos Martín from the University of Alcalá de Henares

The main objective of this study is to analyze the effects on sleep quality and student performance through the application of non-invasive neuromodulation NESA.

The information collected on the academic stress questionnaire at the university, the scale for coping with academic stress and the questionnaire on sociodemographic variables, will be strictly necessary for the purpose indicated in the object of the study and will be treated in accordance with the Regulations. General (EU) 2016/679, on data protection and Organic Law 3/2018, on Personal Data Protection and guarantee of digital rights, with the different universities participating in this clinical trial being responsible for the treatment.

You can exercise the rights: access, rectification, opposition, deletion, portability and limitation to treatment by sending a communication, motivated and accredited, to <a href="mailto:lopd@uax.es">lopd@uax.es</a>. You can also file a claim with the competent Authority in (<a href="mailto:www.aepd.es">www.aepd.es</a>)

This information will not be used for any other purpose outside of this research nor will it be disclosed to third parties.

For more information about the processing of your data, you can contact the UAX Data Protection Officer (<a href="mailto:dpd@uax.es">dpd@uax.es</a>).

The general results of this study can be requested by the participants when it has been completed.



## Based on the above:

- 1. I confirm that I have read and understood the information for the project / research. I have had the opportunity to consider the information, ask questions, and receive satisfactory answers.
- 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without any type of dental care or legal rights being affected.
- 3. I understand that the relevant data collected during the project / research may be used by the researchers of this study for research and subsequent publications.
- 4. Questions related to your participation in this study can be directed to Dr. Pablo Aparicio Montero, with email paparmon@uax.es.

For all these reasons, you expressly consent to the processing of personal data for the indicated purposes.

In Madrid to \_\_\_/ \_\_/ 2 0 \_\_\_

Participant name: -----
Firm:

In the event that the participant is between 12 and 16 years old, I understand all the information collected above and I consent to the processing of the minor's data, as father / mother or legal guardian.

\*Mother's name:

Firm

\*Father's name:

Firm

Firm

Guardian's name:

<sup>\*</sup> The signature of both spouses is required in the case of separated / divorced parents